CLINICAL TRIAL: NCT05321212
Title: Efficacy (Systemic and Cerebral) and Safety of PEMbrolizumab PD-L1-positive (More Than 50% of Tumor Cells), Advanced Non-small-cell Lung Cancer : A Study of Real Life in Brittany .
Brief Title: Efficacy and Safety of PEMbrolizumab PD-L1-positive (>50% of Tumor Cells), Advanced NSCL Cancer(PEMBREIZH)
Acronym: PEMBREIZH
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: PEMBREIZH (29BRC18.0260)
Record Dates: First submitted 2019-08-07; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Immunotherapy
Keywords: pembrolizumab; first line treatment; PDL1 TPS > 50%; brain efficacy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study was a French multicentric cross-sectional study retrospectively of 108 consecutive advanced NSCLC patients with a PD-L1 TPS ≥50% and without EGFR/ALK aberrations treated by pembrolizumab in first line.

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically confirmed NSCLC PD- L1 TPS ≥ 50% stage III and IV WHO performance status of 0, 1 or 2 adequate organ function

Exclusion Criteria:

* previous EGFR or ALK aberrations positive test for hepatitis B or C virus indicating acute or chronic infection known history of testing positive for human immunodeficiency virus (HIV) severe, uncontrolled autoimmune disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Non-small-cell lung cancer with PDL1 TPS > 50% treated in first line with pembrolizumab
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-01-02 (Actual); Study Completion 2019-03-02 (Actual)

PRIMARY OUTCOMES:
progression free survival with pembrolizumab | time from initiation of pembrolizumab to the date of disease progression or death ( 20 months)
  time from initiation of pembrolizumab to the date of disease progression or death

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHRU de Brest, Brest
  - CHIC de QUIMPER, Quimper

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning one year and ending five years following the publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.